CLINICAL TRIAL: NCT02059252
Title: Proof of Concept Study Assessing Safety, Tolerability and Performance of SmartMatrix Dermal Replacement Scaffold
Brief Title: Safety, Tolerability and Performance of SmartMatrix Dermal Replacement Scaffold
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Mode of application to be reconsidered by Sponsor
Sponsor: Smart Matrix Limited (Other)
Collaborators: Welsh Centre for Burns and Plastic Surgery, Swansea, UK (Unknown); Queen Victoria Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SML001/13
Record Dates: First submitted 2013-12-11; First posted 2014-02-11 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-04

CONDITIONS: Basal Cell Carcinoma; Squamous Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SmartMatrix scaffold (Experimental): SmartMatrix dermal replacement scaffold
  Interventions: Device: SmartMatrix dermal replacement scaffold

INTERVENTIONS:
Device: SmartMatrix dermal replacement scaffold — SmartMatrix dermal replacement scaffold

SUMMARY:
SmartMatrix™ is a single layer dermal replacement scaffold for full thickness skin replacement. The scaffold consists of a porous matrix of cross-linked human fibrin plus alginate that has been designed and optimised to facilitate wound closure and healing through cellular ingress and rapid growth of new blood vessels.

This proof of concept study will involve patients with surgical wounds resulting from the excision of basal cell carcinoma (BCC) and squamous cell carcinoma SCC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age
* Suspected or histologically proven BCC or SCC
* Suspected or histologically proven BCC or SCC ≥1cm ≤3cm in diameter on either leg
* Expected defect following surgery ≥3cm, ≤6cm in diameter
* Patient or authorised representative able to comprehend and sign the Informed Consent prior to enrolment in the study

Exclusion Criteria:

* Aged <18 years of age
* Pregnant or lactating females
* Skin lesion >4cm in diameter or size that will result in post-surgical defect >6cm in diameter
* Lesion located over joint, i.e. ankle or knee
* Patient who are smokers
* Diabetic patients
* Patients diagnosed with peripheral vascular disease or venous stasis
* Patients receiving regular systemic steroids
* Patients who are immuno-compromised (either acquired or congenital)
* Patients with a known coagulopathy (either acquired or congenital) but not including patients on aspirin or other anti-platelet therapy
* Patients who have received radiotherapy treatment to the area about to be treated with Smart Matrix
* Concurrent participation in another experimental intervention or drug study
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Safety | 6 months
  incidence of adverse events related to use of wound scaffold

SECONDARY OUTCOMES:
wound healing | 6 months, 12 months
  measurement of time to 100% re-epithelialisation of wound
cosmesis | 6 months, 12 months
  patient and surgeon assessment of scar formation and development using recognised assessment scores
pain at dressing change | 3 months
  pain at dressing change will be assessed using a 10cm VAS
dressing change | 3 months
  frequency and number of dressing changes will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Iain Whitaker, Professor, Principal Investigator — The Welsh Centre for Burns and Plastic Surgery, Morriston Hospital, Swansea, UK
Locations (2):
- United Kingdom (2):
  - Queen Victoria Hospital NHS Foundation Trust, East Grinstead
  - The Welsh Centre for Burns and Plastic Surgery, Swansea